CLINICAL TRIAL: NCT05797376
Title: Effects of aSPIrin Versus Aspirin Plus Low-dose RIvaroxaban on Carotid aTherosclerotic Plaque Inflammation
Acronym: SPIRIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Seung-Whan Lee, M.D., Ph.D., Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-1322
Record Dates: First submitted 2023-03-09; First posted 2023-04-04 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Atherosclerosis of Artery; Coronary Artery Disease; Peripheral Arterial Disease; Carotid Stenosis
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease; Carotid Stenosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban + Aspirin group (Experimental): patients are prescribed aspirin at a daily dose of 100mg and Rivaroxaban (2.5 mg twice a day)
  Interventions: Drug: Rivaroxaban 2.5mg
- Aspirin group (No Intervention): patients are prescribed aspirin at a daily dose of 100mg

INTERVENTIONS:
Drug: Rivaroxaban 2.5mg — patients are prescribed aspirin at a daily dose of 100mg and Rivaroxaban (2.5 mg twice a day)
  Other Names: Xarelto 2.5mg
  Arms: Rivaroxaban + Aspirin group

SUMMARY:
Primary Study Objective : To compare the effects of low-dose rivaroxaban plus aspirin versus aspirin on atherosclerotic plaque inflammation using serial FDG Positron Emission Tomography/Computed Tomography(PET-CT) imaging of carotid artery and ascending aorta.

Secondary Study Objective : To compare the effects of low-dose rivaroxaban plus aspirin versus aspirin on biomarkers including high-sensitivity C-Reactive Protein(CRP) and lipid profiles.

DETAILED DESCRIPTION:
Cardiovascular disease is a major health problem across the world. The age-adjusted death rate for cardiovascular disease has significantly decreased during recent decades, and this decline is related to the widespread use of evidence-based medicines. However, even upon optimal medical therapies, patients remains at a substantial residual risk for acute coronary syndrome (ACS) or acute ischemic stroke(AIS), requiring new therapeutic approaches. Plaque rupture and subsequent thrombus formation is the most common cause of ACS and AIS. Atherosclerosis is a chronic immune-inflammatory disorder. Inflammation is believed to be critically important to plaque rupture by destroying the fibrous cap, thereby predisposing to ACS and AIS. Cross-talk between coagulation and inflammatory pathway via protease-activated receptor (PAR) activation has been recognized . Factor Xa is responsible for promoting inflammation, which participate in the atherosclerotic process and plaque destabilization either directly via activation of PARs or indirectly through the generation of thrombin .

In the Cardiovascular Outcomes for People Using Anticoagulation Strategies (COMPASS) trial, the rate of a composite of cardiovascular death, stroke, or myocardial infarction was lower by 24% with low-dose rivaroxaban (2.5 mg twice daily) plus aspirin than with aspirin alone among patients with stable atherosclerotic vascular disease, but the rate of major bleeding was higher by 70%. Interestingly, the rate of stroke was remarkably lower by 42% with rivaroxaban plus aspirin than with aspirin alone. The substantial net clinical benefits seen with rivaroxaban plus aspirin may not be fully explained by their anti-thrombotic effect alone, suggesting pleiotropic effects coupled with factor Xa antagonism. Besides its role in hemostasis and thrombosis, low-dose rivaroxaban may inhibit atherosclerotic plaque inflammation and decrease plaque destabilization. To test this hypothesis, the investigators will compare the effects of aspirin versus aspirin plus low-dose rivaroxaban on carotid atherosclerotic plaque inflammation using serial 18F-fluorodeoxyglucose (FDG) Positron Emission Tomography/Computed Tomography(PET-CT) imaging of carotid artery and ascending aorta.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age inclusive
* Asymptomatic Carotid Artery Disease (diameter stenosis, 20-80%)
* Inclusion criteria for the COMPASS trial (stable Peripheral Artery Disease(PAD); or stable Coronary Artery Disease(CAD) with 1 of age over 65 years, or age <65 years plus atherosclerosis less than 2 vascular beds or less than 2 additional risk factors)
* FDG Postron Emission Tomography(PET)/Computed tomogrphy(CT) shows hot uptakes at carotid artery (with or without hot uptake at ascending aorta)
* The patient or guardian agrees to the study protocol and the schedule of clinical and FDG Postron Emission Tomography(PET)/Computed tomogrphy(CT) follow-up, and provides informed, written consent, as approved by the Institutional Review Board/Ethical Committee.

Exclusion Criteria:

* Patients treated with carotid endarterectomy or stent placement
* Contraindications to rivaroxaban or aspirin.
* Stroke in 1 month or any hemorrhagic or lacuna stroke
* Need for dual antiplatelet therapy or oral anticoagulant therapy
* Severe left ventricular dysfunction (ejection fraction < 30%)
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (alanine aminotransferase(ALT) or aspartate aminotransferase(AST) > 3 times upper limit of normal).
* Unwillingness or inability to comply with the procedures described in this protocol.
* Patient's pregnant or breast-feeding or child-bearing potential.
* Insulin requiring diabetes
* Patients who have experienced critical organ bleeding within 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
The percent change (%) in Most Diseased segment(MDS) Target-to-Background Ratio(TBR) of the index vessel | 12 months
  The percent change (%) in Most Diseased segment(MDS) Target-to-Background Ratio(TBR) of the index vessel defined as (Most Diseased segment(MDS) Target-to-Background Ratio(TBR) at 12 months - Most Diseased segment(MDS) Target-to-Background Ratio(TBR) at baseline)/(Most Diseased segment(MDS) Target-to-Background Ratio(TBR) at baseline)*100.
  * Index vessel: carotid artery with the highest 18-FDG uptake at baseline

SECONDARY OUTCOMES:
Change from baseline in whole vessel Target-to-Background Ratio(TBR) | 12 months
  Change from baseline in whole vessel Target-to-Background Ratio(TBR) within the index vessel, Most Diseased segment(MDS) Target-to-Background Ratio(TBR), & whole vessel Target-to-Background Ratio(TBR) of the aorta.
Change from baseline in hs-C-Ractive Protein(CRP) and lipid profiles | 12 months
  Change from baseline in hs-C Ractive Protein(CRP) in mg/dL and lipid profiles(total cholesterol in mg/dL, Triglyceride(TG) in mg/dL, High Density Lipoprotein(HDL) in mg/dL, Low Density Lipoprotein(LDL) in mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No